CLINICAL TRIAL: NCT05584956
Title: Clinical Study to Evaluate the Possible Efficacy and Safety of L- Carnitine and Sildenafil in Children Having Beta Thalassemia With Increased Tricuspid Regurgitant Jet Velocity
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Zaki Zedan, Clinical pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beta thalassemia
Record Dates: First submitted 2022-10-13; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Beta Thalassemia With Increased Tricuspid Regurgitant Jet Velocity
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): n=22): Patients will receive traditional treatment and L- carnitine 50mg/kg/day orally (maximum dose 3g per day)
  Interventions: Drug: L_carnitine
- Group 2 (Active Comparator): n=22): Patients will receive traditional treatment and Sildenafil 0.25mg/kg/dose every 6 h orally (maximum dose 60 mg per day)
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: L_carnitine — l-carnitine stabilizes red blood cell membranes and thus improves the anemic state[
  Arms: Group 1
Drug: Sildenafil — selective and potent inhibitor of cGMP-specific phosphodiesterase 5 (PDE5), which promotes smooth muscle relaxation in lung vasculature, has been used successfully in the treatment of primary and secondary PH.
  Arms: Group 2

SUMMARY:
This study aims to investigate the possible efficacy and safety of L_Carnitine and Sildenafil on patient with Beta thalassemia complicated with increased Tricuspid Regurgitant Jet Velocity

ELIGIBILITY:
Inclusion Criteria:

* Children with Beta thalassemia major who have increased TRJV more than 2.5m/s.
* Children age from 6-18 years

Exclusion Criteria:

* Others hemolytic anemia

  * Young age before 6 years of age
  * Allergy to Sildenafil or L-carnitine
  * Patient with documented causes of pulmonary hypertension rather than caused by Beta thalassemia.
  * Hepatic dysfunction: serum Alanine Aminotransferase (ALT) 3X.
  * Renal dysfunction: Creatinine level greater than or equal to 1.2 mg/dl.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-07-08 (Estimated); Study Completion 2024-07-08 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary functions | 3 months
  change in the studied cardiopulmonary functions at the baseline and 3 months after intervention

SECONDARY OUTCOMES:
Biochemical parameters | 3 months
  Changes in Vascular Endothelial Growth Factor level (VEGF) at baseline and 3 months after the intervention
Biochemical parameters | 3 months
  Changes in Nitric oxide level (NO) at the baseline and 3 months after the intervention
Biochemical parameters | 3 months
  Changes in ferritin serum level at the baseline and 3 months after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Kamal Hegazy, Professor, Principal Investigator — Tanta University
Locations (1):
- Tanta University Hospital, Tanta, Gharbia Governorate, Egypt